CLINICAL TRIAL: NCT05828615
Title: Effects of Breathing Control vs Alternate Nostril Breathing on Maternal Cardiovascular Parameters in Pregnancy Induced Hypertension
Brief Title: Breathing Exercise in Pregnancy-induced Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Rec/01385 Rida Kanwal
Record Dates: First submitted 2023-04-12; First posted 2023-04-25 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Pregnancy Induced Hypertension
Keywords: Breathing control; Alternate nostril breathing; Maternal cardiovascular parameters; Fetal Heart rate
MeSH Terms: conditions — Hypertension, Pregnancy-Induced

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Alternate nostril breathing exercise 2 times a day, 10 min duration of exercise each time, for 5 days
  Interventions: Other: Group A
- Group B (Active Comparator): Breathing control exercise 2 times a day, 10 min duration of exercise each time, for 5 days
  Interventions: Other: Group B

INTERVENTIONS:
Other: Group A — Close your eyes and exhale through your left nostril fully and slowly, once you have exhaled completely, release your right nostril and place your ring finger on the left nostril.
  Breathe in deeply and slowly from the right side. Make sure your breath is smooth and continuous. Aerobics exercises (Walking): 3-5 days per week at moderate intensity, of approximately 30 minutes.
  Start slowly and gradually increase your walking pace over 3 minutes until the activity feels moderate (slightly increased breathing, but should still be able to talk.
  Walk at a moderate pace for about 10 minutes the first then gradually increase time with RPE(8-9).
  Other Names: Alternate nostril breathing
  Arms: Group A
Other: Group B — The position of the woman should be relaxed and comfortable e.g., crock lying, sitting, standing position. Place one hand on chest and other on stomach and close eyes to relax and focus on breathing. Slowly breathe in through nose with your closed mouth.Breathe out through your nose and try to use as small effort as possible and make your breaths slow, relaxed and smooth.
  Aerobics exercises (Walking): 3-5 days per week at moderate intensity, of approximately 30 minutes.
  Start slowly and gradually increase your walking pace over 3 minutes until the activity feels moderate (slightly increased breathing, but should still be able to talk.
  Walk at a moderate pace for about 10 minutes the first then gradually increase time with RPE(8-9).
  Arms: Group B

SUMMARY:
To determine the effects of Breathing control vs Alternate nostril breathing on maternal cardiovascular parameters in pregnancy and to determine the effect of breathing control vs Alternate nostril breathing on Fetal Heart rate. Many evidence-based studies show breathing exercises have beneficial and useful effects on the hypertensive population and also have positive effects on pregnancy-induced hypertension.

DETAILED DESCRIPTION:
Many breathing interventions are used for pregnancy-induced hypertension but the comparison is limited between two breathing techniques. In this study, a comparison will be carried out between evidence-based breathing techniques including breathing control and alternate nostril breathing to see which of these two exercises gives the best effects on females with pregnancy-induced hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Females with 3rd-trimester pregnancies included
* BMI<3
* Diagnosed pregnancy-induced HTN

Exclusion Criteria:

* An exaggerated response to exercise on BP ( 160/110 mmHg )
* Uncontrolled Diabetics or asthma
* Cardiac diseases
* Orthopedic complications
* Using anti-epileptic drugs and
* Hyperthyroidism or hypothyroidism

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 46 (Actual)
Dates: Start 2023-04-10 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Blood Pressure | 12 weeks
  Changes from baseline to 4 weeks after the intervention, time of discharge from the hospital, and, 40 days postpartum, measured through a sphygmomanometer. Blood pressure is measured in millimeters of mercury (mm Hg). A blood pressure measurement has two numbers Systolic and Diastolic. The patients are classified according to the range as follows. Hypertension stage 1 SYSTOLIC (mm of Hg): 131-139, DIASTOLIC (mm of Hg): 81-89 and stage 2 SYSTOLIC (mm of Hg): 140 and above, DIASTOLIC (mm of Hg): 90 and above
Oxygen Saturation | 12 weeks
  Changes from baseline to 4 weeks after the intervention, time of discharge from the hospital, and, 40 days postpartum, measured through a pulse oximeter. It measures how much oxygen is in person's blood. It is a small device, clips onto a finger, earlobe or another part of the body. Oxygen saturation level of 95% is considered typical for most healthy people, a level of 92% or lower can indicate potential hypoxemia, which is a seriously low level of oxygen in the blood.
Functional capacity | 12 weeks
  Changes from baseline to 4 weeks after the intervention, and, 40 days postpartum, measured through 6 min walk test (6 MWT) used to measure Functional capacity. It is a submaximal exercise test that can aid in assessing the functional capacity of patients with cardiopulmonary diseases, in this test we find out the maximum distance in meters that an individual covers in 6 min without any support.
Quality of life(QOL) (postpartum) | 12 weeks
  Changes from baseline to 4 weeks after intervention and 40 days postpartum measured through Short Form 36 Health Survey Questionnaire (SF-36) that is used to indicate the health status of particular population. Its consists of eight scaled scores, which are weighted sums of the questions in each section. Each scale is directly transformed into a 0-100 scale on assumption that every question carries equal weight and lower score the more disability.

SECONDARY OUTCOMES:
Fetal Heart rate | 8 weeks
  Changes from baseline to Changes from baseline to 4 weeks after intervention and time of delivery measured through Doppler ultrasound (US).This is a method that uses a device to listen and record heartbeat of baby through abdomen. The rate and pattern of heart rate of baby shown on a screen and printed on paper. The average fetal heart rate is between 110 and 160 beats per minute.

CONTACTS AND LOCATIONS:
Overall Officials: Mehwish Waseem, MSPT(CPPT), Principal Investigator — Riphah International University
Locations (1):
- Punjab medical center Gujarat., Dhok Gujra, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aalami M, Jafarnejad F, ModarresGharavi M. The effects of progressive muscular relaxation and breathing control technique on blood pressure during pregnancy. Iran J Nurs Midwifery Res. 2016 May-Jun;21(3):331-6. doi: 10.4103/1735-9066.180382. PMID 27186213
- [Background] Felton M, Hundley VA, Grigsby S, McConnell AK. Effects of slow and deep breathing on reducing obstetric intervention in women with pregnancy-induced hypertension: a feasibility study protocol. Hypertens Pregnancy. 2021 Feb;40(1):81-87. doi: 10.1080/10641955.2020.1869250. Epub 2021 Jan 19. PMID 33463384
- [Background] Tsakiridis I, Bakaloudi DR, Oikonomidou AC, Dagklis T, Chourdakis M. Exercise during pregnancy: a comparative review of guidelines. J Perinat Med. 2020 Jul 28;48(6):519-525. doi: 10.1515/jpm-2019-0419. PMID 32619194